CLINICAL TRIAL: NCT00677937
Title: A Randomised Controlled Trial to Investigate an Educational Programme and Continuous Monitoring to Prevent Diabetes in Individuals With Screen Detected Pre-diabetes in a Multi-ethnic Population
Brief Title: A Diabetes Prevention Study Targeting High Risk Individuals With Education and Ongoing Support
Acronym: PREVENTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UHL10564
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes mellitus; prevention; education; impaired glucose tolerance; multi-ethnic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intervention to include education and ongoing support
  Interventions: Behavioral: Modified DESMOND education and ongoing support
- 2 (No Intervention): Control to receive standard care

INTERVENTIONS:
Behavioral: Modified DESMOND education and ongoing support — 6 hours of education with 1 month of inclusion, 3 years of ongoing support including annual refresher sessions
  Arms: 1

SUMMARY:
The study aims to identify people at high diabetes risk within the local population and then implement and evaluate a pragmatic and low-cost diabetes prevention programme containing structured education on lifestyle, physical activity and food choices. An ongoing support framework will continue to reinforce and maintain the participant's individual goals to prevent the development of diabetes and reduce cardiovascular risk.

Therefore the principal question is: can we significantly reduce the incidence of diabetes through structured education in a high risk multi-ethnic UK population?

DETAILED DESCRIPTION:
T2DM is an increasing chronic disease affecting over 2 million people in England alone, shortens life and consumes 10% of NHS resources. At diagnosis many have established complications involving damage to the eyes, kidneys, feet and heart. There is a need to focus efforts to prevent this devastating disease. One in 7 adults have Pre-diabetes (PDM) with 50% developing T2DM over the next 5-10 years. There is clear evidence that treating subjects with PDM with an intensive lifestyle modification programme (LSMP) dramatically reduces T2DM. These programmes are not cost effective, involve intensive use of resources and are unproven in the UK. Some minority ethnic groups have a higher risk of T2DM, any LSMP would need to be culturally sensitive. Our objective is to test if we can develop a low cost but effective LSMP for the UK. We will develop a training programme to skill healthcare professionals and non-professionals and so called 'lay' educators to deliver the LSMP. Benefits of lay educators are patient involvement in a patient centred service and the contribution to building capacity within the NHS workforce. We will develop a simple self-assessment tool to identify those at highest risk of T2DM. We will conduct a clinical trial, testing the LSMP in 50 practices and 816 patients. The practices will be randomised to either a control or intervention 'arm'. Control practices will give information to patients at risk in line with current best practice. Subjects in the Intervention practices will be invited to the LSMP and will receive 6 hours of group education over 3 months plus ongoing contact. Subjects will be followed for 3 years. The LSMP will encourage individuals to scrutinise information, ask questions, and self-manage their condition, using simple, non-technical language and visual aids. This approach has been effective in T2DM and we will use this model along with expertise in physical activity and lifestyle change, working with leading experts. The study is designed to show if we can significantly reduce the risk of developing T2DM, as well as the effect on weight, blood pressure, patients' quality of life, physical activity and dietary behaviours. We will demonstrate its cost effectiveness to ensure relevance to the NHS. The research team have international expertise in prevention of T2DM.

ELIGIBILITY:
Patients that will be included into the study if they have either / or

* Diagnosed with Pre-Diabetes (IGT or IFG)
* Aged 40 - 75 if English speaking European or 25 - 75 if South Asian
* Able to attend group education sessions

Exclusion Criteria:

Patients will be excluded from the study if they are:

* Unable to give consent
* Unable to attend group education sessions
* Diagnosis of diabetes at screening or during the study
* Require an interpreter for language other than South Asian

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2009-05; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Reduction in incidence of diabetes at 3 years | 3 years from entry into the study

SECONDARY OUTCOMES:
change in hba1c, fasting and post glucose levels, cardiovascular risk (framingham), presence of MetS (NCEP ATP III) | 3 years from enrollment into the study

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Davies, MD, FRCP, Principal Investigator — University Hospitals, Leicester; Kamlesh Khunti, Principal Investigator — Univeristy of Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Yates T, Gray LJ, Henson J, Edwardson CL, Khunti K, Davies MJ. Impact of Depression and Anxiety on Change to Physical Activity Following a Pragmatic Diabetes Prevention Program Within Primary Care: Pooled Analysis From Two Randomized Controlled Trials. Diabetes Care. 2019 Oct;42(10):1847-1853. doi: 10.2337/dc19-0400. Epub 2019 Aug 9. PMID 31399440
- [Derived] Yates T, Henson J, Edwardson C, Bodicoat DH, Davies MJ, Khunti K. Differences in levels of physical activity between White and South Asian populations within a healthcare setting: impact of measurement type in a cross-sectional study. BMJ Open. 2015 Jul 23;5(7):e006181. doi: 10.1136/bmjopen-2014-006181. PMID 26204908
- [Derived] Bodicoat DH, O'Donovan G, Dalton AM, Gray LJ, Yates T, Edwardson C, Hill S, Webb DR, Khunti K, Davies MJ, Jones AP. The association between neighbourhood greenspace and type 2 diabetes in a large cross-sectional study. BMJ Open. 2014 Dec 23;4(12):e006076. doi: 10.1136/bmjopen-2014-006076. PMID 25537783
- [Derived] Gray LJ, Khunti K, Williams S, Goldby S, Troughton J, Yates T, Gray A, Davies MJ; Let's Prevent Collaborators. Let's prevent diabetes: study protocol for a cluster randomised controlled trial of an educational intervention in a multi-ethnic UK population with screen detected impaired glucose regulation. Cardiovasc Diabetol. 2012 May 20;11:56. doi: 10.1186/1475-2840-11-56. PMID 22607160
- See also: in-dept diabetes information site from University Hospitals of Leicester — http://www.leicestershirediabetes.org.uk/353.html